CLINICAL TRIAL: NCT06009198
Title: Nutritional, Water, Sanitation and Hygiene Related Education Intervention to Address Malnutrition of Early Adolescents in Pakistan: A School Based Study: Protocol
Brief Title: Nutritional, and WASH Related Education Intervention to Address Malnutrition of Early Adolescents in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Rozina Karmaliani, Dr, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: : 2021-3572-19378
Record Dates: First submitted 2022-09-16; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Malnutrition
Keywords: Adolescents; Nutrition; School; Body Mass Index; WASH
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance Education with Iron Folate Supplement (Experimental): 1. Nutrition education
  2. WASH education
  3. Micronutrient supplementation
  Interventions: Drug: Iron folate tablets
- Routine Education (No Intervention): Routine school education

INTERVENTIONS:
Drug: Iron folate tablets — Iron folate tablets will be administered to the underweight school going adolescents girls and boys to see the affect on BMI and micronutrients
  Other Names: Nutrition and WASH education
  Arms: Advance Education with Iron Folate Supplement

SUMMARY:
Globally, one of the major risk factor for adolescent's morbidity is considered Malnutrition. Worldwide adolescent age group 10-19 is increasing and they are at increased risk of malnutrition related diseases resulting in high morbidity and mortality. Asian countries are suffering with the double burden of malnutrition including Pakistan. The risk factors that contribute to malnutrition in the population includes unsafe drinking water, poor sanitary conditions, lack of proper waste disposal facilities, poor health awareness, poor nutrition and hygiene. However, studies have shown that nutrition education, and water, sanitation, hygiene (WASH) programmes in the schools are effective strategies to promote the health status of the adolescents (girls and boys). The primary objective of this study is to determine a school based nutrition and WASH education intervention to improve nutritional status among early adolescents.

DETAILED DESCRIPTION:
This study is a Cluster Randomized Control Trial. Two stage sampling technique will be done. The sample size was calculated by using PASS software. Sample sizes was estimated to change in nutritional status of the early adolescent boys and girls. Sample size of 360 adolescents (180 in each intervention and control group) will achieve 80% power assuming 42% malnutrition among students in control arm and at least 6% reduction in the intervention arm having 90 students from each school at a two-sided 5% level of significance.

To assess the micronutrient levels (Iron, Zinc, Calcium, Complete Blood Count ) through blood sample, a subset of 108 adolescents 6-8 grade school going adolescents (54 intervention group,54 control group) from this total sample size (360) will be selected through random selection.

Data will be collected through adopted and adapted self-administered, structured questionnaire from 6,7, and 8 grade school going adolescents at base line and at end line.

To approach to 6, 7, and 8 grade adolescents, informed consent will be first taken from their mothers/immediate caretaker and school management. Before collecting the data, a written informed assent will also be taken from the participants available in Urdu and . Study participants will be briefed about purpose of the study and assured about anonymity and confidentiality of information shared. Finally, the survey questionnaire will be completed . In case, participants have any queries related to the questionnaire, explanation will be provided to them. Physical assessment will be done by the principal investigator which will take almost 10 minutes/ individual. For the biochemical markers assistance from local Aga Khan Laboratory will be sought. Phlebotomist /lab assistance from Aga Khan laboratory will go to the concerned educational institute and draw blood samples from the participants who have given their consent for the test.

Data analysis plan Quantitative variables will be described by means and standard deviations whereas median with interquartile range will be mentioned for qualitative variables. Frequencies and percentages will be calculated for knowledge, attitude and practices of adolescents regarding nutrition and WASH. The comparison between intervention and control at base line and end line will be performed by using paired t-test and Chi-square. For the variables that are not normally distributed, nonparametric test McNamara will be used. Binary logistic regression and multiple linear regression will be used to assess the effect of intervention. All the statistical analysis will be conducted using SPSS version 23. P value less than 0.05 will be considered statistically significant.

Intervention will be planned on the basis of socio ecological model and health promoting school framework. School health environment, health education, health services and nutrition programs will be focused in the intervention stage of the study .

Sixteen sessions (one session per week) will be arranged on nutrition education and water, sanitation, and hygiene for adolescents. Micronutrient tablets will be administered to the adolescents for three months on daily basis through school teachers. In addition, Cooking recipe in local language will be shared with adolescent's mother/immediate care takers through adolescents.

During the intervention phase, there is no such risks involve to the study participants except their valuable time. Due to micronutrient supplementation there may be temporary dizziness,nausea,headache, constipation, and dark color stool along with discomfort from prick for blood drawing from adolescents. To reduce the temporary side effects of administration of micronutrients , researcher will advise them to keep adequately hydrated themselves and take the micronutrients supplementation tablet during meal. Reassurance regarding drawing the blood samples will be done. Existing referral system will be identified and utilized if needed Study Approval will be obtained from the Aga khan University Ethical Review Committee (ERC). Approval will also be sort from the participating school management in Gojra. Any identification information like name and personnel information will be replaced by codes to address anonymity issue. Confidentiality of the data will be ensured by keeping the data under safe custody, electronic files will also be password protected. Only the primary investigator will access the raw data and the research team members involved in data analysis. Respect for human dignity will be safeguarded by completely informing the participants about all aspects of the study including purpose, their rights including right to withdraw from the study at any point, and all possible risks and benefits. This information will be communicated verbally as well as in writing in the form of consent /assent. For the adolescent's participation, assent will be obtained after taking permission from their parents / immediate caretaker.

Trial will be conducted in compliance with the protocol, Good Clinical Practice and the applicable regulatory requirement(s).

ELIGIBILITY:
Inclusion Criteria:

* All students studying in 6, 7, and 8 grade
* Informed consent given by adolescent's mothers/immediate care takers
* Assent given by the adolescent at baseline

Exclusion Criteria:

* Students leave the school during study • Consent not given by the mother/immediate care taker will be excluded from the analysis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 635 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Knowledge regarding nutrition and WASH | 16 weeks
  knowledge of adolescents will be assessed by employing adapted tool from the FAO publication Guidelines which was developed by the Food and agriculture organization of the united nations. It is an extract from the FAO publication Guidelines for assessing nutrition-related Knowledge, attitudes, and practices (2014), also called KAP manual and it is available at http://www.fao.org/docrep/019/i3545e/i3545e00.htm
  The knowledge part comprises 16 questions, each question with multiple options to assess the knowledge regarding food items, their consumption, and their effect on the health of adolescents. The knowledge will be assessed before and after intervention for comparison.
Attitude regarding nutrition and WASH | 16 weeks
  Attitude of adolescents will be assessed by employing adapted tool from the FAO publication Guidelines which was developed by the Food and agriculture organization of the united nations. it is an extract from the FAO publication Guidelines for assessing nutrition-related knowledge, attitudes and practices (2014), also called KAP manual and it is available at http://www.fao.org/docrep/019/i3545e/i3545e00.htm The attitude part covers 5 questions to know the perceived benefits and perceived barriers regarding food consumption before and after the intervention
Practices regarding nutrition and WASH | 16 weeks
  Practices of adolescents will be assessed by employing adapted tool from the FAO publication Guidelines which was developed by the Food and agriculture organization of the united nations. it is an extract from the FAO publication Guidelines for assessing nutrition-related Knowledge, attitudes, and Practices (2014), also called the KAP manual and it is available at http://www.fao.org/docrep/019/i3545e/i3545e00.htm The practices part contains 11 questions that address the practices regarding the consumption of food and behaviors. Pre and Post-intervention assessment of practices will evaluate the efficacy of the education sessions.

SECONDARY OUTCOMES:
Body Mass Index | 16 weeks
  According to the Centre for Disease Control, guidelines will be followed to calculate Body Mass Index. Initially, the height and weight of all participants will be measured. the BMI will be calculated on the age parameter. This will help in determining a person's health on the basis of being Underweight, normal, Overweight, and obese. The criteria are as follow:
  BMI Categories:
  Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9 Obesity = BMI of 30 or greater

OTHER OUTCOMES:
Changes in Symptoms of malnutrition and micronutrient status | 16 weeks
  A complete blood picture and blood level of calcium and Zinc will be measured prior to the intervention to gather baseline data. the blood test will be repeated 04 weeks after the intervention implementation. The changes in level will be compared and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Rozina Karmaliani, Dr, Principal Investigator — Aga Khan University school of Nursing and Midwifery karachi,pakistan
Locations (1):
- Aga Khan University karachi,pakistan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data is shared on the whole through publication. The individual data will not be shared with any researcher The study findings will also shared with stake holders

DOCUMENTS (1):
  • Study Protocol (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT06009198/Prot_000.pdf